CLINICAL TRIAL: NCT03060343
Title: Preliminary Clinical Study of Autologous T Cells Modified Chimeric Antigen Receptor (CAR) Targeting PD-L1 and CD80/CD86 (Zeushield Cytotoxic T Lymphocytes) for the Treatment of Recurrent or Refractory Non Small Cell Lung Cancer
Brief Title: Zeushield Cytotoxic T Lymphocytes (Z-CTLs) for Relapsed or Refractory Non Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu Fenglei (Other)
Collaborators: Hunan Zhaotai Yongren Medical Innovation Co. Ltd. (Other); Hunan Yongren Medical Innovation Co. Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Yu Fenglei, Chief of the Thoracic Surgery Department, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z-NSCLC-01
Record Dates: First submitted 2017-02-12; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zeushield Cytotoxic T Lymphocytes (Experimental): Enrolled patients will receive Zeushield Cytotoxic T Lymphocytes by infusion
  Interventions: Biological: Zeushield Cytotoxic T Lymphocytes

INTERVENTIONS:
Biological: Zeushield Cytotoxic T Lymphocytes — Three dose levels will be evaluated. Dose Level One: 1.0×10^5 cells/kg, Dose Level Two: 1.0×10^6 cells/kg, Dose Level Three: 1.0×10^7 cells/kg.
  At the discretion of the investigator, if patients with active disease have stable disease or a response at week 8 or on subsequent evaluations, they are eligible to receive up to 6 additional infusions at 8 to 12 week intervals.

SUMMARY:
A single-center, open-label pilot study to determine the safety, tolerance and engraftment potential of zeushield cytotoxic T lymphocytes in subjects with PD-L1+ positive non-small cell lung cancer.

DETAILED DESCRIPTION:
The purpose of this first in human study is to determine the safety and feasibility of Zeushield Cytotoxic T Lymphocytes(Z-CTLs) in patients with relapsed or refractory NSCLC. Z-CTLs therapy is a novel immunotherapy under investigation in which patients have their T-cells (a type of white blood cell) collected and modified in the laboratory, before they are given back to the patient. The T-cells are modified to transform the intracellular signal domain of PD-1 and CTLA-4 to immune activation stimulus signal and transform T cells to a new kind of cancer-killer cells: zeushield cytotoxic T lymphocytes (Z-CTls).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged >18 years old
* Subjects are diagnosed as refractory, recurrent ,metastatic, advanced non-small cell lung cancer by histological and cytological methods including specific lesion-targeted brush biopsy, lavage and fine needle aspiration;
* Have at least one new measurable tumor lesion compared with previous irradiated region
* Tumor tissues samples confirmed as PD-L1 positive
* Expected survival≥12 weeks
* ECOG scored as 0-1 or KPS grading > 80
* PLT≥100000/mm3
* Hb≥9.0g/dL
* Serum creatinine≤2.5mg/dL，CCR≥50ml/min (renal malfunction defined as CCR<50ml/min according to Cockroft-Gault formula)
* ALT and AST≤2.5ULN; for liver metastasis，ALT and AST ≤5ULN
* Serum TBiL≤3.0mg/dL, TBiL≤2.5ULN
* PT: INR < 1.7 or extended PT to normal value < 4s
* Adequate venous access for apheresis or venous blood collection, and no other contraindication of blood cell separation
* Patients with willingness to be in this study and able to provide informed consent
* Capable of receiving treatment and follow up, included subjects are required to receive treatment in the enrolled centre
* Women of childbearing age are required to take acceptable measures to minimize the possibility of pregnancy during whole session. Women of childbearing age must have negative results of serum or urine tests within 24 hours prior to infusion. Women subjects must not be in lactation;

Exclusion Criteria:

* pregnant women or women in lactation
* active HBV or HCV infection
* HIV/AIDS infection
* active infection
* previously suffered from diseases or concurrent diseases as followed：
* patients confirmed as severe autoimmune diseases in long-term (over 2 months) need of systemic immune inhibitors (steroid) or as immune-mediated symptomatic diseases including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune vasculitis (for example, Wegener's granulomatosis)
* subjects with previous diagnosis as motor neurone disease caused by autoimmunity
* subjects previously suffered from toxic epidermal necrolysis (TEN)
* subjects with any mental diseases including dementia, mental status change that may impinge the understanding and performance of informed consent and related questionnaire
* subjects with severe, uncontrollable diseases judged by investigators that may hinder them receiving this treatment
* subjects with previously active malignant tumors including basal or squamous skin cancer, superficial bladder cancer, and in situ breast carcinoma within 5 years who had been completely cured without the need of follow-up treatment are not excluded.
* during ongoing treatment using systemic steroid or steroid inhalants
* subjects with unstable or active peptic ulcer or alimentary tract hemorrhage
* subjects with previous organ transplantation or ready for organ transplantation
* subjects in need of anticoagulant therapy treatment (warfarin or heparin)
* subjects judged by investigators as not appropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-11-28 (Estimated); Study Completion 2019-11-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 8 weeks
  Observe and determine the potential adverse events related to the escalating dose infusion of Z-CTLs such as high fever,jaundice, kidney failure and so on.

SECONDARY OUTCOMES:
Number of Z-CTLs in peripheral blood samples after infusion | 8 weeks
  Detect Z-CTLs in peripheral blood samples after infusion by flow cytometry every week
Objective response rate (ORR) | 2 years
  the ratio of patients diagnosed as partial remission (PR) to complete remission (CR) according to RECIST 1.1 criteria
Progression free survival (PFS) | 2 years
  the duration from baseline to PD (audited and confirmed by independent imaging), or to the day of any death event
Time to tumor progression (TTP) | 2 years
  the duration from baseline to disease starts to get worse or spreads to other parts of the body
Overall survival (OS) | 2 years
  the time period from the 1st day of treatment to the day of death for any reason. For patients who are still alive at the data analysis day, OS data is subject to the last confirmed time of survival patients

CONTACTS AND LOCATIONS:
Overall Officials: Yu Fenglei, MD, PhD, Principal Investigator — Second Xiangya Hospital of Central South University; Li Peng, PhD, Principal Investigator — Hunan Zhaotai Yongren Medical Innovation Co. Ltd.
Locations (1):
- Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided